CLINICAL TRIAL: NCT01833377
Title: Caraway Intake as a Sustainable Dietary Practice: Impact on Overweight & Obese Women
Brief Title: Effect of Consumption of Caraway on Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT12345678
Record Dates: First submitted 2013-03-26; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight; BMI
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- caraway sample (Experimental): caraway sample
  Interventions: Dietary Supplement: caraway sample
- Placebo (Active Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: caraway sample
  Other Names: caraway water extract product
  Arms: caraway sample
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the applicability of caraway (black cumin) intake on the treatment of obesity. So, a randomized placebo controlled clinical trial will be conducted to examine the applicability of caraway product in terms of safety and efficacy.

DETAILED DESCRIPTION:
A randomized placebo-controlled clinical trial, was done on 120 healthy overweight and obese women aged 20-55 in Iran. data were collected trough questionaires, interview and physical examination. the required parameters including anthropometric indices, body composition vital parameters (heart rate and blood pressure)and full blood parameters, were measured before and after intervention. volunteers were randomized into test and control group and were asked to consume either caraway samples or placebo during 12 intervention weeks.

the outcome measure will be assessed for both primary and secondary data from baseline through week 12 (3 months).

ELIGIBILITY:
Inclusion Criteria:

* overweight and obese women (BMI> 25)
* aged 20-55 years old
* healthy subjects

Exclusion Criteria:

* Pregnant and lactating women
* Thyroid disease
* type I or II diabetes mellitus
* hypertension (systolic BP 140 and/or diastolic BP 90)
* endocrine dysfunction
* impaired liver function
* chronic renal disease
* cardiovascular disease
* primary dyslipidemia
* myopathy
* patients using drugs which affect on metabolism or appetite
* a maintained weight loss in the preceding 3 months
* meals not eaten at regular intervals
* participation in another investigation study within the past 30 days
* a history of alcohol or drug abuse within the past year
* smoking
* a history of sleep disorders
* clinical depression or other psychiatric conditions
* abnormal obese
* allergy or sensitivity to any of the 'active' or 'placebo' product ingredients

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | Baseline and 12 weeks
  The changes in BMI from baseline at 12 weeks are measured.

SECONDARY OUTCOMES:
change in all blood parameters | Baseline and 12 weeks
  The changes in all blood parameters from baseline at 12 weeks are measured.
Change in vital parameters (systolic and diastolic blood pressure and pulse rate) | Baseline and 12 weeks
  The changes in systolic and diastolic blood pressure and pulse rate from baseline at 12 weeks are measured.
Change in body weight | Baseline and 12 weeks
  The changes in body weight from baseline at 12 weeks are measured.
Change in anthropometric indices including waist, hip, thigh and mid-upper arm circumference (cm) | Baseline and 12 weeks
  The changes in anthropometric indices including waist, hip, thigh and mid-upper arm circumference from baseline at 12 weeks are measured.
Change in appetite | Baseline and 12 weeks
  The changes in appetite from baseline at 12 weeks are measured.
Change in body composition including fat percentage, muscle mass, lean body mass, bone mass and water percentage | Baseline and 12 weeks
  The changes in body composition from baseline at 12 weeks are measured.
Change in body weight (kg) | Baseline and 12 weeks
  The changes in body weight from baseline at 12 weeks are measured.
Change in basic and active metabolic rate | Baseline and 12 weeks
  The changes in BMR and AMR from baseline at 12 weeks are measured.
Change in food intake | Baseline and 12 weeks
  Change in food intake
  The changes in food intake (macro and micro nutrient intake) from baseline at 12 weeks are measured.
Change in urine specific gravity | Baseline and 12 weeks
  The changes in urine specific gravity from baseline at 12 weeks are measured.

CONTACTS AND LOCATIONS:
Overall Officials: che wan jasimah mohamed radzi, PhD, Study Chair — University of Malaya; Majid Hajifaraji, PhD, Study Director — Shahid Beheshti University of Medical Sciences

REFERENCES:
- [Derived] Kazemipoor M, Rezaeian M, Kazemipoor M, Hamzah S, Shandilya SK. Computational Intelligence Techniques for Assessing Anthropometric Indices Changes in Female Athletes. Curr Med Imaging. 2020;16(4):288-295. doi: 10.2174/1573405614666180905111814. PMID 32410532
- [Derived] Kazemipoor M, Radzi CW, Hajifaraji M, Haerian BS, Mosaddegh MH, Cordell GA. Antiobesity effect of caraway extract on overweight and obese women: a randomized, triple-blind, placebo-controlled clinical trial. Evid Based Complement Alternat Med. 2013;2013:928582. doi: 10.1155/2013/928582. Epub 2013 Nov 10. PMID 24319489